CLINICAL TRIAL: NCT04477889
Title: Methodist Health System COVID-19 Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 024.CRI.2020.A
Record Dates: First submitted 2020-07-17; First posted 2020-07-20 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Cohort: Patients treated at MHS facilites for COVID-19
  Interventions: Other: Treatment for COVID-19
- Synopsis for COVID Bariatric, Hepato-Biliary and Colorectal surgery study: 30 Day Mortality after surgery in patients with COVID19 infection who undergo elective bariatric, hepato-biliary and colorectal surgery.
  * Patients diagnosed with COVID-19 at the time of surgery up to seven days before surgery
  * Patients diagnosed with COVID-19 within 30 days after surgery
  Interventions: Other: Treatment for COVID-19

INTERVENTIONS:
Other: Treatment for COVID-19 — Patients treated for COVID-19

SUMMARY:
This is a prospective cohort observational registry study that will include data on all patients who are treated at MHS facilities for COVID-19.

DETAILED DESCRIPTION:
This is a prospective cohort observational registry study that will include data on all patients who are treated at MHS facilities for COVID-19. Data including, but not limited to demographics, comorbidities, medications, treatment, and clinical outcomes will be collected from February 2020 to December 2025. Subjects will undergo no additional tests or procedures as part of this registry study. All patient data will be obtained from the patient's electronic health records (EHR) of the hospital or clinic in a retrospective manner. The process for gathering the data will not influence treatment decisions. There will be no direct patient contact associated with inclusion in this registry study.

ELIGIBILITY:
Inclusion Criteria:

* Patient tested positive for COVID-19 (SARS-CoV-2)
* Patient sought care for COVID-19 at a MHS facility
* Aged 18 years or older

Exclusion Criteria:

* Patient that do not have COVID-19
* Non-confirmed COVID-19 patients
* Aged 17 years or younger

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients who are treated at MHS facilities for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient Characteristics | June 2020 - Dec 2025
  Patient characteristics
Treatment Measures and Intervention strategies | June 2020 - Dec 2025
  Treatment measures and intervention strategies
Clinical and survival outcomes | June 2020 - Dec 2025
  Clinical and survival outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Crystee Cooper, DHEd, Principal Investigator — Methodist Health System
Locations (1):
- Clinical Research Institute Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No